CLINICAL TRIAL: NCT02580578
Title: A Multicentre Prospective Non-interventional Study Assessing the Management of Canadian Women With Uterine Fibroids, a Patient Registry
Brief Title: A Multicenter Prospective Non-Interventional Study Assessing the Management of Canadian Women With Uterine Fibroids
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMO-CAN-WH-0412
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Leiomyoma
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Female patients who are diagnosed and treated for symptoms associated with their uterine fibroids per routine clinical practice. No intervention is administered in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention is administered in this study.

SUMMARY:
This study will characterize the treatments and outcomes associated with different uterine fibroid treatments in Canada, to understand patients' preferences and satisfaction with different medical and procedural interventions. The study will also assess the effectiveness of ulipristal acetate (Fibristal®) in controlling bleeding, reducing fibroid volume and symptoms, and improvement in patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

-Pre-menopausal adult women with confirmed diagnosis and symptoms associated with uterine fibroids who are initiating treatment.

Exclusion Criteria:

-Significant pelvic pathology not associated with uterine fibroids.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with uterine fibroids treated as per standard of care in clinical practice.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Uterine Fibroid Symptom Quality of Life 37-Item Questionnaire (UFS QoL) | 24 Months
Ruta Menorrhagia (Bleeding) 15-Item Questionnaire | 24 Months
Number of Participants with Adverse Drug Reactions | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Enciu, Study Director — Allergan
Locations (20):
- Canada (20):
  - Peter Lougheed Centre/University of Calgary, Calgary, Alberta
  - Urestky Edmonton Clinic, Edmonton, Alberta
  - Sanders Vancouver Clinic, Vancouver, British Columbia
  - Children's and Women's Health Centre of British Columbia - The University of British Columbia, Vancouver, British Columbia
  - Southern Health Centre, White Rock, British Columbia
  - Landau Fredericton Clinic, Fredericton, New Brunswick
  - Strand Clinic, St. John's, Newfoundland and Labrador
  - IWK Healtch Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Minimally Invasive Gynecology Clinic, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - St. Micheals Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - South Windsor Women's Health, Windsor, Ontario
  - Centre Gynécologie et Maternité, LaSalle, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Clinique de Gynécologie & Obstétrique Pierre Boucher, Montreal, Quebec
  - Complexe Medical Saint-Laurent, Saint-Laurent, Quebec
  - University of Saskatchewan, Regina, Saskatchewan
  - CHU de Québec-Universite Laval, Québec

REFERENCES:
- [Derived] Bougie O, Bedaiwy MA, Laberge P, Lebovic G, Leyland N, Atri M, Murji A; CAPTURE Steering Committee. Quality of ultrasonography reporting and factors associated with selection of imaging modality for uterine fibroids in Canada: results from a prospective cohort registry. CMAJ Open. 2020 Aug 12;8(3):E506-E513. doi: 10.9778/cmajo.20200004. Print 2020 Jul-Sep. PMID 32792350
- [Derived] Bedaiwy MA, Janiszewski P, Singh SS; CAPTURE Steering Committee. A Patient Registry for the Management of Uterine Fibroids in Canada: Protocol for a Multicenter, Prospective, Noninterventional Study. JMIR Res Protoc. 2018 Nov 20;7(11):e10926. doi: 10.2196/10926. PMID 30459144